CLINICAL TRIAL: NCT02497547
Title: A Phase 2b, Double-blind, Randomized, Parallel, Placebo-Controlled, Multiple-Dose Study to Evaluate the 12-week Efficacy of Vagitocin in Postmenopausal Women With Symptoms of Vaginal Atrophy
Brief Title: An Efficacy Study of Vagitocin in Postmenopausal Women With Symptoms of Vaginal Atrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PepTonic Medical AB (Industry)
Collaborators: A+ Science AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXYPEP201
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Atrophy
Keywords: Atrophy; Pathological Conditions, Anatomical; Oxytocin; Oxytocics
MeSH Terms: conditions — Atrophy; Pathological Conditions, Anatomical | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oxytocin 400 IU (Experimental): Oxytocin 400 IU vaginal gel (1 x 1mL/400 IU oxytocin daily for 12 weeks)
  Interventions: Drug: Oxytocin
- Oxytocin 200 IU (Experimental): Oxytocin 200 IU vaginal gel (1 x 1mL/200 IU oxytocin daily for 12 weeks)
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo vaginal gel (1 x 1mL daily for 12 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin
  Other Names: Vagitocin
  Arms: Oxytocin 200 IU; Oxytocin 400 IU
Drug: Placebo
  Arms: Placebo

SUMMARY:
Up to 50% of postmenopausal women frequently suffer from atrophic vaginitis or vaginal atrophy with symptoms including vaginal dryness, irritation, burning, itching or discomfort. Vaginal atrophy is a consequence of the lining tissue of the vagina becoming thinner, drier, and less elastic due to lack of estrogen. In addition, vaginal atrophy is associated with an increased pH, which creates an environment more susceptible to infections.

Menopausal hormone therapy is a common treatment for vaginal atrophy. However, menopausal hormone therapy has been shown to coincide with an increased incidence of breast cancer, heart attack and stroke. Some women experience adverse reactions such as uterine bleeding, perineal pain, and breast pain with menopausal hormone therapy. Many women are also reluctant to initiate estrogen treatment, due to a general negative view of menopausal hormone therapy in the society. There are also many contraindicated conditions like undiagnosed vaginal bleeding, thromboembolic disease, breast cancer, other estrogen-sensitive cancers, or liver disease. Women suffering from vaginal atrophy and presenting with these conditions have extremely limited options for effective therapy.

Oxytocin is a peptide hormone, normally released into the circulation via the pituitary. Oxytocin has been shown in vitro to exert positive effects on the proliferation of human vaginal mucosal cells from postmenopausal women. Local application of oxytocin, in the form of a vaginal gel, Vagitocin, has been investigated in previous studies on postmenopausal women, as a new effective and safe option for the treatment of vaginal atrophy. Vagitocin appeared to reverse the manifestation of vaginal atrophy by stimulating vaginal mucosal growth, reducing symptoms of vaginal atrophy and increasing the patients' wellbeing and quality of life. Overall, treatment with Vagitocin was safe and well tolerated by the subjects in the studies.

In this study, the clinical efficacy of Vagitocin as a potential treatment for postmenopausal women suffering from moderate to severe symptoms of vaginal atrophy, vaginal irritation/itching and vaginal discomfort and/or pain associated with sexual activity will be explored. In addition, the dose relationship and lowest effective dose of Vagitocin will be investigated.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, a subject must:

1. Be a female subject between the ages of 40 and 65 years at the time of randomization, who is willing to participate in the study as indicated by signing the informed consent
2. Be a postmenopausal woman with at least 24 months of spontaneous amenorrhea or a woman, who has had surgical bilateral oophorectomy with or without hysterectomy at least 6 weeks ago
3. Have ≤ 5% superficial cells in vaginal smear cytology at screening
4. Have a vaginal pH > 5.0 at screening
5. Have a level of estradiol ≤ 30 pg/mL and a level of Follicle Stimulating Hormone (FSH) > 40 milli International Units (mIU)/ml at screening
6. Have one moderate to severe vaginal atrophy symptom (vaginal irritation and itching, dyspareunia, vaginal dryness, dysuria or presence of vaginal bleeding associated with sexual activity) that has been identified by the subject as being the most bothersome to her
7. Have a Body Mass Index (BMI) ≤32 kg/m2
8. Be judged by the Principal Investigator or Sub-investigator as being in otherwise good health based on a pre-study medical evaluation performed within 35 days prior to the initial dose of study medication
9. Have endometrial thickness of < 4 mm as determined by vaginal ultrasonography, in women with an intact uterus
10. Be willing to abstain from sexual activity and the use of vaginal douching within 24 hours prior to vaginal pH measurements at screening and at Visits 2 and 3

Exclusion Criteria:

To participate in the study, a subject must not:

1. Be currently hospitalized
2. Have a history of ongoing cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychological, or musculoskeletal disease or disorder that is clinically significant in the opinion of the Principal Investigator or Sub-Investigator
3. Have had or have any known or suspected tumor disease that is clinically significant in the opinion of the Principal Investigator or Sub-Investigator
4. Have a history of endometrial hyperplasia or uterine/endometrial, breast or ovarian cancer
5. Have a history of undiagnosed vaginal bleeding
6. Have an ongoing urogenital infection at randomization visit
7. Any contraindication to oxytocin therapy and allergy to the use of oxytocin and any components of the investigational drugs
8. Have a history of drug and/or alcohol abuse within one year of start of study
9. Have used any prescription or Over The Counter (OTC) medications including phytoestrogens, herbal medicinal products or hormonal intra-uterine device with known estrogenic effects within 12 weeks prior to screening procedures
10. Have used any type of vaginal lubricants and moisturizers within 24 hours prior to screening procedures
11. Have used estrogen alone or estrogen/progestin for any of the time periods specified in the protocol
12. Have any reason, which in the opinion of the Principal Investigator or Sub-Investigator would prevent the subject from safely participating in the study or complying with protocol requirements
13. Have participated in another clinical trial within 90 days prior to screening, have received an investigational drug within the three months prior to the initial dose of study medication, or be likely to participate in a clinical trial or receive another investigational medication during the study
14. Have contraindication to any planned study procedure

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 12 in severity of vaginal atrophy symptom that has been self-identified by the subject as being the most bothersome to her in the vaginal atrophy questionnaire | After 12 weeks of treatment
  Vaginal atrophy symptoms: vaginal irritation and itching, dyspareunia, vaginal dryness, dysuria or presence of vaginal bleeding associated with sexual activity
Change from baseline to Week 12 in % superficial cells (increase is positive) | After 12 weeks of treatment
Change from baseline to Week 12 in Vaginal pH (decrease is positive) | After 12 weeks of treatment

SECONDARY OUTCOMES:
Change from baseline to Week 4 in severity of the vaginal atrophy symptoms that has been self-identified by the subject as being the most bothersome to her in the vaginal atrophy questionnaire | After 4 weeks of treatment
  Vaginal atrophy symptoms: vaginal irritation and itching, dyspareunia, vaginal dryness, dysuria and the absence or presence of vaginal bleeding associated with sexual activity
Change from baseline to Week 4 in % superficial cells (increase is positive) | After 4 weeks of treatment
Change from baseline to Week 4 in vaginal pH (decrease is positive) | After 4 weeks of treatment
Change from baseline to week 4 and 12 of % parabasal cells (decrease is positive) | After 4 and 12 weeks of treatment
Change from baseline to week 4 and 12 of maturation value (increase is positive) | After 4 and 12 weeks of treatment
Change from baseline to Weeks 4 and 12 in severity of vaginal atrophy symptoms self-assessed by the subject in the vaginal atrophy questionnaire | After 4 and 12 weeks of treatment
  Vaginal atrophy symtoms: vulvar and vaginal irritation and itching, dyspareunia, vaginal dryness, dysuria and the absence or presence of vaginal bleeding associated with sexual activity
Change from baseline to Week 12 in Quality of Life evaluation parameters | After 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Aino F Jonasson, MD, Principal Investigator — Karolinska Universitetssjukhuset, Huddinge
Locations (5):
- Sweden (5):
  - Hoftekliniken, Helsingborg
  - Qvinnolivet Specialistläkarna Kungsbacka, Kungsbacka
  - Kvinnoforskningsenheten, Karolinska Universitetssjukhuset, Huddinge, Stockholm
  - Kvinnokliniken, Norrlands Universitetssjukhus, Umeå
  - Kvinnokliniken, Akademiska sjukhuset, Uppsala